CLINICAL TRIAL: NCT02273076
Title: Predicting Breast Flap Necrosis by Spatial Frequency Domain Imaging
Status: Withdrawn | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Gregory Evans, M.D., Chair, Department of Plastic Surgery, University of California, Irvine
Other Study IDs: 20141229
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Disorders of Skin Grafts and Flaps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Spatial Frequency Domain Imaging — Spatial Frequency Domain Imaging

SUMMARY:
The current surgical procedure for breast diseases places an emphasis on the conservation of breast skin in order to provide more optimal reconstruction.

The purpose of this study is to use portable, non-contact optical imaging device developed at the Beckman Laser Institute called Spatial Frequency Domain Imaging to detect the changes in a skin during reconstructive surgery procedure and healing process.

DETAILED DESCRIPTION:
The researchers can use Spatial Frequency Domain Imaging instrument to measure the concentration of blood flow in the skin tissue and can determine of the changes that observed in the properties of the mastectomy flap that may be delay in healing process.

The imaging device can determine the change from baseline measurement to the development of skin necrosis, wound infection, or implant extrusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female 18 years and older scheduled for breast reconstructive surgery.

Exclusion Criteria:

* Minor and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population will be recruited from UCI Anesthetic and Plastic Surgery Institute clinics, seen by the Plastic Surgery Service. Subjects requiring breast reconstructive surgery using either implant based or autologous reconstruction will be identified.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
skin flap healing | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Evans, MD, Principal Investigator — UCIMC
Locations (1):
- UCIMC, Orange, California, United States